CLINICAL TRIAL: NCT04176549
Title: The Assessment of Biomarkers in Ectopic Pregnancy
Brief Title: Assessment of Biomarkers in Ectopic Pregnancy
Acronym: AMBER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4883
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Ectopic Pregnancy
Keywords: Ectopic Pregnancy; Biomarker
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples Serum samples Urine samples Oral swabs Vaginal swabs Fallopian tube samples Peritoneal washing samples Trophoblast tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ectopic Pregnancy: Patients diagnosed with ectopic pregnancy Samples collected: Plasma, Serum, Urine, Oral swab, Vaginal Swab If surgery required for tubal ectopic: Fallopian tube, peritoneal washing, trophoblast
  Interventions: Other: Management of Ectopic Pregnancy
- Surgical termination of pregnancy: Patients undergoing elective surgical termination of pregnancy Samples collected: Plasma, Serum, Urine, Oral swab Vaginal swab, Trophoblast
  Interventions: Other: Management of termination of pregnancy
- Elective hysterectomy and salpingo-oophorectomy: Patients undergoing elective hysterectomy and salpingo-oophorectomy Samples collected: Fallopian tube, peritoneal washing
  Interventions: Other: Elective management of gynaecology patients

INTERVENTIONS:
Other: Management of Ectopic Pregnancy — Expectant, Medical or Surgical management of Ectopic Pregnancy
  Groups: Ectopic Pregnancy
Other: Management of termination of pregnancy — Surgical termination of pregnancy
  Groups: Surgical termination of pregnancy
Other: Elective management of gynaecology patients — Elective hysterectomy and salpingo-oophorectomy
  Groups: Elective hysterectomy and salpingo-oophorectomy

SUMMARY:
To further develop a patient care pathway (incorporating a statistical model which uses the values of biomarkers) in routine clinical practice that will aid the diagnosis and management of women with an ectopic pregnancy.

DETAILED DESCRIPTION:
Purpose and design-There is a need for the patient care pathway to evolve in order to aid and improve the diagnosis and management of women with a pregnancy of unknown location (PUL) and ectopic pregnancy (EP). There is potential for this to be achieved by the incorporation of a statistical model that uses one or more novel markers identified by this study. These markers may replace or add to the effectiveness of markers used in the current statistical model.

Recruitment-200 patients. Inclusion: Patients attending the Early Pregnancy Unit (EPU) in the first trimester with a PUL or ectopic pregnancy on trans-vaginal ultrasound scan between the ages of 18-50 years. Exclusion: Patients diagnosed with cancer, presence of acute medical condition, patients aged less than 18 years, patients who cannot give fully informed study consent.

Consent - Posters will advertise the study. Patients in EPU will be invited to the study by a member of the clinical care team. Written consent will be required for all aspects of the study other than for 3-dimensional scanning of PUL and EP patients, where verbal consent will be obtained. Patients will be given at least 24 hours to consider whether they wish to participate.

Confidentiality - The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act. Patient consent forms will be stored securely within the study file. All patient identifiable information, where required, will be stored electronically on National Health Service (NHS) approved computers, accessible only by personnel involved in the study via password.

Conflict of interest - None involved in the study have a conflict of interest.

Dissemination of results - No patient identifiable information will be included in the research report or publication. Anonymised results will be disseminated to scientific community by means of publication in peer-reviewed literature and presented at national and international meetings.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Early Pregnancy Unit (EPU) in the first trimester (up to 14 weeks gestation) with a PUL or ectopic pregnancy on trans-vaginal ultrasound scan between the ages of 18 and 50 years.
* Patients attending the gynaecology unit for a surgical termination of pregnancy or for a salpingo-oophorectomy.

Exclusion Criteria:

* Patients diagnosed with cancer, presence of an acute medical condition, patients aged less than 18 years, patients who cannot give fully informed study consent (language or learning impairment), presence of a viable intrauterine pregnancy and presence of miscarriage.
* Exclusion to fallopian tube samples - presence of any ectopic pregnancy that does not require operative salpingectomy.
* Exclusion to peritoneal washings - presence of any ectopic pregnancy that does not require access to the peritoneal cavity as part of management.
* Exclusion to trophoblast tissue sampling - presence of an ectopic pregnancy that does not require surgical removal.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Pregnant women attending the Early Pregnancy Unit (EPU) within a hospital in the first trimester (up to 14 weeks gestation) with a PUL or ectopic pregnancy on trans-vaginal ultrasound scan between the ages of 18 and 50 years.
  * Women attending the gynaecology unit for a surgical termination of pregnancy or for a salpingo-oophorectomy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Novel biomarkers for Ectopic Pregnancy prediction and diagnosis | 3 years
  Identification of microRNA and microbiome markers identified in blood, urine, swabs, fallopian tubes, peritoneal washings and trophoblastic tissue that have predictive value in identifying ectopic pregnancies as well as high and low risk pregnancy of unknown location. microRNA will be assessed using blood and trophoblast using cell free profiling assays and quantitative reverse transcription polymerase chain reaction and microbiome will be assessed using Illumina microbiome genomic sequencing.

SECONDARY OUTCOMES:
microRNA as a biomarker | 3 years
  Identification of novel microRNA markers from blood and trophoblast tissue samples associated with ectopic pregnancy and high-risk pregnancy of unknown location. MicroRNA will be assessed using blood and trophoblast using cell free profiling assays and quantitative reverse transcription polymerase chain reaction.
Microbiome as a biomarker | 3 years
  Identification of novel microbiome markers from blood and trophoblast tissue samples associated with ectopic pregnancy and high-risk pregnancy of unknown location. Microbiome will be assessed using Illumina microbiome genomic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bourne, MBBS, PhD, MRCOG, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bobdiwala S, Al-Memar M, Farren J, Bourne T. Factors to consider in pregnancy of unknown location. Womens Health (Lond). 2017 Aug;13(2):27-33. doi: 10.1177/1745505717709677. Epub 2017 Jun 29. PMID 28660799
- [Background] Senapati S, Barnhart KT. Biomarkers for ectopic pregnancy and pregnancy of unknown location. Fertil Steril. 2013 Mar 15;99(4):1107-16. doi: 10.1016/j.fertnstert.2012.11.038. Epub 2013 Jan 3. PMID 23290746
- [Background] Van Calster B, Bobdiwala S, Guha S, Van Hoorde K, Al-Memar M, Harvey R, Farren J, Kirk E, Condous G, Sur S, Stalder C, Timmerman D, Bourne T. Managing pregnancy of unknown location based on initial serum progesterone and serial serum hCG levels: development and validation of a two-step triage protocol. Ultrasound Obstet Gynecol. 2016 Nov;48(5):642-649. doi: 10.1002/uog.15864. Epub 2016 Oct 9. PMID 26776599
- [Background] Bobdiwala S, Christodoulou E, Farren J, Mitchell-Jones N, Kyriacou C, Al-Memar M, Ayim F, Chohan B, Kirk E, Abughazza O, Guruwadahyarhalli B, Guha S, Vathanan V, Bottomley C, Gould D, Stalder C, Timmerman D, van Calster B, Bourne T. Triaging women with pregnancy of unknown location using two-step protocol including M6 model: clinical implementation study. Ultrasound Obstet Gynecol. 2020 Jan;55(1):105-114. doi: 10.1002/uog.20420. PMID 31385381
- [Background] Cook J, Bennett PR, Kim SH, Teoh TG, Sykes L, Kindinger LM, Garrett A, Binkhamis R, MacIntyre DA, Terzidou V. First Trimester Circulating MicroRNA Biomarkers Predictive of Subsequent Preterm Delivery and Cervical Shortening. Sci Rep. 2019 Apr 10;9(1):5861. doi: 10.1038/s41598-019-42166-1. PMID 30971726